CLINICAL TRIAL: NCT01440166
Title: A Single Center, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of CAT-1004 in Healthy Adult Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of CAT-1004 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CAT-1004-101
Record Dates: First submitted 2011-09-08; First posted 2011-09-26 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Human healthy volunteers
MeSH Terms: interventions — Pharmaceutical Preparations; edasalonexent

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1 / Dose level 1 (Experimental): Single dose orally: CAT-1004 Dose level 1 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 2 / Dose level 2 (Experimental): Single dose orally: CAT-1004 Dose level 2 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 3 /Dose level 3 (Experimental): Single dose orally: CAT-1004 Dose level 3 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 4/ Dose level 4 (Experimental): Single dose orally: CAT-1004 Dose level 4 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 5/ Dose level 5 (Experimental): Single dose orally: CAT-1004 Dose level 5 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 2/ Dose level 2 ( FE) (Experimental): Single dose orally (Under fed conditions): CAT-1004 Dose level 2 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 3/ Dose level 3 (FE) (Experimental): Single dose orally (Under fed conditions): CAT-1004 Dose level 3 or placebo
  Interventions: Drug: Drug; Other: Placebo
- Cohort 6 / Dose level 6 (FE) (Experimental): Single dose orally (Under fed conditions) CAT-1004 Dose level 4 or placebo Subjects may be reenrolled from Cohort 4.
  Interventions: Drug: Drug; Other: Placebo
- Cohort 7 / Dose level 7 (FE) (Experimental): Single dose orally (Under fed conditions)CAT-1004 Dose level 5 or placebo Subjects may be reenrolled from Cohort 5.
  Interventions: Drug: Drug; Other: Placebo

INTERVENTIONS:
Drug: Drug — Single dose oral administration of CAT1004 or placebo-6 to 8 subjects will be treated with CAT-1004 per cohort.
  Other Names: CAT-1004
Other: Placebo — Single dose oral administration of CAT1004 or placebo- 2 subjects treated with placebo per cohort.

SUMMARY:
* To evaluate the safety and tolerability of escalating single doses of CAT-1004 relative to placebo in healthy adult volunteers.
* To evaluate the pharmacokinetics (PK) of escalating single doses of CAT-1004 in healthy adult volunteers.
* To evaluate the effect of a high-fat meal on single doses of CAT-1004 in healthy adult volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. In good health.
2. Age: 19 to 55 years inclusive at Screening.
3. Satisfies one of the following

   * Females not of childbearing potential: non-pregnant and non-lactating; surgically sterile or postmenopausal, OR
   * Males: surgically sterile, abstinent, or subject or partner is utilizing an acceptable contraceptive method during and 3 months after the last study dose.
4. BMI: 18 to 30 kg/m2 at Screening.

Key Exclusion Criteria:

1. Clinically significant abnormalities in physical examination or vital signs.
2. Clinically significant electrocardiogram (ECG) abnormalities as assessed by the investigator.
3. Clinically significant screening laboratory result as assessed by the Investigator.
4. The subject has a history of clinically significant allergies (except for untreated, asymptomatic seasonal allergies at the time of dosing), or hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
5. History or presence of malignancy with the past 5 years.
6. History of alcohol or substance abuse or eating disorder within 2 years, OR regular use of alcohol within 6 months (>14 units of alcohol per week; 1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
7. Use of any investigational drug or participation in any investigational study within 30 days prior to screening. For dose levels 6 and 7 fed cohorts, subjects may participate who have taken part in the dose levels 4 and 5 fasted cohort.
8. Any significant blood loss within 60 days prior to screening, e.g. blood donation, participation in study with multiple blood draws, etc.
9. Any condition, disease, disorder or clinically relevant laboratory abnormality that, in the opinion of the Investigator, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment.
10. A suspected allergy or sensitivity to CAT-1004 or excipients based upon known allergies to excipients or compounds of a similar class.
11. Any clinically significant systemic infection within 3 weeks prior to screening.
12. Use of prescription medications within 30 days of screening.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety | Change from Baseline versus Day-1 though 72 hrs post dose and EOT/FU
  Safety Endpoints: Laboratory evaluations including hematology, chemistry, coagulation and urinalysis, physical examinations, AEs, serious AEs (SAEs), ECGs, and vital signs.

SECONDARY OUTCOMES:
Pharmacokinetic Profile | Plasma blood samples through 72 hrs, urine collections through 48 hrs
  The following noncompartmental PK parameters will be calculated: area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf), area under concentration-time curve from time 0 to time of last quantifiable concentration (AUClast), maximum observed plasma concentration (Cmax), time to first occurrence of Cmax (Tmax), terminal phase elimination half-life (t½), apparent oral clearance (CL/F), and volume of distribution during the terminal phase (Vz/F). Additional PK parameters may be calculated if deemed appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Clinical Research Unit, Lincoln, Nebraska, United States